CLINICAL TRIAL: NCT06116994
Title: The Effect of Using Camouflaged Dental Syringe on Children's Anxiety and Behavioral Pain
Brief Title: The Effect of Using Camouflaged Dental Syringe
Acronym: Camouflage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Sara Mustafa Bagher, Associate Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 053-02-19
Record Dates: First submitted 2023-10-23; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Anxiety, Dental; Behavior
Keywords: Alligator syringe sleeve; anxiety; buccal infiltration; camouflaged syringe; local anesthesia; pediatric dentistry
MeSH Terms: conditions — Anxiety Disorders; Behavior

STUDY DESIGN:
Intervention Model Description: Case Control
Who Masked: Outcomes Assessor
Masking Description: Impossibility to blind the participant and operator to the intervention. The statistician was blinded to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): In the control group, subjects will receive the buccal infiltration anesthesia using the traditional dental syringe.
  Interventions: Other: The buccal infiltration anesthesia with a conventional dental syringe
- Test group (Experimental): Subjects in the test group will receive the buccal infiltration anesthesia with the camouflaged dental syringe.
  Interventions: Other: The buccal infiltration anesthesia with a camouflaged dental syringe (Angelus ™)

INTERVENTIONS:
Other: The buccal infiltration anesthesia with a camouflaged dental syringe (Angelus ™) — In the test group, subjects will receive buccal infiltration anesthesia with the a camouflaged dental syringe. The used camouflaged dental syringe (Angelus ™) will consist of an alligator-shaped syringe sleeve that covers the dental syringe and makes it more friendly without affecting its function. The alligator-shaped syringe sleeve has three main components, which are the mouth, trunk, and rear feet. The mouth of the alligator sleeve covers the local anesthesia needle, the trunk covers the syringe barrel of the traditional dental syringe, and the rear feet hold the finger grip.
  Arms: Test group
Other: The buccal infiltration anesthesia with a conventional dental syringe — In the control group, subjects will receive buccal infiltration anesthesia with the conventional dental syringe.
  Arms: control group

SUMMARY:
Seeing the dental syringe can be terrifying, especially for young children. Hiding the dental syringe during local anesthesia (LA) administration can sometimes be challenging for the pediatric dentist. Therefore, this randomized clinical trial aims to assess the effect of a camouflaged dental syringe on children's anxiety and behavioral pain in comparison to the traditional dental syringe during local anesthesia administration in pediatric patients. It will include cooperative and healthy 6-10-year-old children scheduled for non-urgent dental treatment that requires buccal infiltration anesthesia (BIA) in the maxillary arch. The subjects will be randomized into either the test or the control groups. In the test group, subjects will receive BIA using the camouflaged dental syringe. Subjects in the control group will receive the BIA using the traditional dental syringe. A single-trained dentist will administer all the anesthesia. Heart rate (HR) will be monitored at three different time points (before, during, and after) the BIA administration. Subjects' anxiety and behavioral pain will be measured through Venham's Anxiety Rating Scale (VARS) and the Face, Leg, Activity, Cry, and Consolability (FLACC) scale, respectively, by two trained and calibrated investigators.

DETAILED DESCRIPTION:
This randomized clinical trial will take place at the Pediatric Dentistry clinics at King Abdulaziz University Faculty of Dentistry (KAUFD). Ethical approval will be obtained from the Research Ethical Committee at King Abdulaziz University (053-02-19).

The dental files of all the children scheduled for non-urgent dental treatment at the Pediatric Dentistry Department clinics during the study period will be reviewed by a single trained general dentist to identify potentially eligible subjects.

Inclusion criteria will include healthy and cooperative 6-10-year-old children with no known allergy and/or sensitivity to local anesthesia and who are scheduled for non-urgent dental treatment that requires buccal infiltration anesthesia (BIA) of at least one maxillary molar.

The cooperation level of the children will be determined based on the child's behavior recorded in the dental file in their previous dental visits. Only children who will be reported to be positive or absolute positive according to Frankel's behavior rating scale will be considered eligible. Children who will be reported to be uncooperative during their previous dental visit or those who did not receive any previous dental treatment at KAUFD and, therefore, have no dental record will be excluded.

The same dentist will approach those who meet the inclusion criteria, and the research aim will be introduced to the legal guardians/parents. An Arabic consent and assent form will be signed by those who agreed to participate.

Before the treatment, subjects will be randomized into a test or control group following a predetermined randomization sequence. In the control group, subjects will receive the BIA using the traditional dental syringe. In contrast, subjects in the test group will receive BIA with the camouflaged dental syringe. The camouflaged dental syringe (Angelus ™) consists of an alligator-shaped syringe sleeve that covers the dental syringe and makes it more friendly without affecting its function. The alligator-shaped syringe sleeve has three main components, which are the mouth, trunk, and rear feet. The mouth of the alligator sleeve covers the LA needle, the trunk covers the syringe barrel of the traditional dental syringe, and the rear feet hold the finger grip. The operator has to place his finger over the rear feet to gain support, then place his thumb inside the thumb ring of the dental syringe to introduce the solution of the local anesthesia.

A single-trained general dentist will give all the injections. All the subjects will be informed that the dentist will give the sleeping juice to help the teeth fall asleep, and the operator in both groups will make sure to keep the needle part of the dental syringe out of the subjects' sight. At the injection site, the oral mucosa will be dried, and topical Benzocaine gel 20% (Sky-Caine Gel, Skydent) will be applied for two minutes. Then, a 30-gauge short needle (Septoject XL, Septodont) will be inserted in the mucobuccal fold without touching the bone. Finally, the needle will be withdrawn. Due to the nature of the study, neither the operator nor the subjects will be blinded to the treatment group.

Heart rate (HR) will be monitored and recorded as beat per minute (bpm) at three-time points: as a baseline before local anesthesia administration, during the needle insertion, and one minute after local anesthesia administration will be completed by using a pulse oximeter (iCare Fingertip Pulse Oximeter, blood oxygen and heartbeats measurement oximeter, OLED screen, White - At101C). In addition, during the administration of the local anesthesia, the subjects will be recorded using a high-resolution camera. Later, two trained and calibrated investigators will watch the videos and evaluate the anxiety level of the subjects using Venham's Anxiety Rating Scale (VARS) and the behavioral pain level using the Face, Leg, Activity, Cry, and Consolability Scale (FLACC). The VARS scores range from zero to five, where zero represents a relaxed, quiet child, and five represents a screaming child. The FLACC scale consists of five categories, each with a score range from zero to two. Moreover, the total scores range from zero to 10, with zero being relaxed and comfortable and 10 being severe discomfort or pain or both.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy
2. Cooperative
3. 6-10-year-old children
4. With no known allergy and/or sensitivity to local anesthesia and who are scheduled for non-urgent dental treatment that requires buccal infiltration anesthesia of at least one maxillary molar

Exclusion Criteria:

1. Children who were reported to be uncooperative during their previous dental visit
2. Children who did not receive any previous dental treatment at KAUFD and, therefore, have no dental record will be excluded.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | at three different time points. As a baseline before Local anesthesia administration, the second will be during the needle insertion, and the third point will be one minute after Local anesthesia administration is completed by using a pulse oximeter
  Heart rate (HR)
Anxiety | during the administration of the local anesthesia, the subjects will be recorded using a high-resolution camera. Later, two trained and calibrated investigators will watch the videos and evaluate the anxiety level of the subjects
  Venham's Anxiety Rating Scale (VARS)
Behavioral pain | during the administration of the local anesthesia, the subjects will be recorded using a high-resolution camera. Later, two trained and calibrated investigators will watch the videos and evaluate the anxiety level of the subjects
  Face, Leg, Activity, Cry, and Consolability Scale (FLACC)

CONTACTS AND LOCATIONS:
Locations (1):
- King AbdulAziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No